CLINICAL TRIAL: NCT07104292
Title: PFMT During Pregnancy - Its Implementation and Effects on Pelvic Floor Disorders, Sexual Function and Obstetric Outcomes: a Hybrid Type 1 Design Randomised Controlled Trial
Brief Title: Pelvic Floor Muscle Training During Pregnancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SHS-KS-06-2025
Record Dates: First submitted 2025-07-10; First posted 2025-08-05 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Pelvic Floor; Urinary Incontinence; Anal Incontinence; Pelvic Organ Prolapse; Sexual Dysfunction
MeSH Terms: conditions — Urinary Incontinence; Encopresis; Pelvic Organ Prolapse; Sexual Dysfunction, Physiological | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic Floor Muscle Training (PFMT) (Experimental): A Danish professional pelvic floor physiotherapist together with a midwife and an urogynecologist have created a free of charge training program, which is easily accessible via a danish website "www.kvindekrop.dk" or via the app "Pelvic FloorTrainer". The women will receive an easily accessible, home-based PFMT program electronically in which they will be motivated to start and engage during pregnancy with continuity after birth.
  Interventions: Behavioral: PFMT
- Standard care (Placebo Comparator): The control group will receive routine care - recommendation to do the training without any further instructions.
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: PFMT — The motivation-informed intervention will tackle both exercise engagement and exercise adherence. Participating women will be introduced to the app and its videos following training. The participants will be introduced not only to muscle training, but also to muscle relaxation. The training will be recommended three to four times a week during pregnancy with further continuity after giving birth.
  Arms: Pelvic Floor Muscle Training (PFMT)
Behavioral: Standard care — Standard care
  Arms: Standard care

SUMMARY:
The project seeks to investigate effectiveness of PFMT during pregnancy.

DETAILED DESCRIPTION:
First-time pregnant women will be recruited through visitations received from family doctors in all obstetrics departments of the Southern Denmark Region. Women will be randomised into two groups: ( Pelvic Floor Muscle Training) PFMT and a control group (standard care). The motivation-informed intervention will tackle both exercise engagement and exercise adherence. The women will receive an easily accessible, home-based PFMT program electronically in which they will be motivated to start and engage during pregnancy with continuity after birth. The data regarding pelvic floor disorders will be obtained at baseline, follow-ups once every trimester of pregnancy, as well as six weeks, three months, and six months postpartum with further follow-up after the study. The data regarding obstetric outcomes will be collected from electronic patient records. For evaluation of implementation process, data regarding motivation and training acceptability will be obtained via questionnaire at the baseline and at follow-up together with telephonically interviews during pregnancy and postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Woman in the 1st trimester of pregnancy (up to 12+6 weeks of gestation)
* Para 0 (no previous birth or pregnancy > 16 weeks of gestation)
* Understands, writes, and reads fluently in Danish or English
* Has a smart phone or computer/tablet to reach the training program

Exclusion Criteria:

* Severe psychiatric illness (e.g. schizophrenia, bipolar disorder, severe depression or anxiety)
* Active substance abuse
* Acute social crises (e.g. homelessness, ongoing domestic violence, severe financial instability, lack of social support)
* Women with limited capacity to provide informed consent (due to cognitive impairment or language barriers)
* Previous pregnancy of > 16 weeks of gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 734 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Urinary incontinence (UI) incidence at 3 months postpartum | At 3 months follow-up after giving birth
  International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) score between 0 (perfect continence) and 21 (total incontinence).

SECONDARY OUTCOMES:
Urinary incontinence at the 1st trimester of pregnancy | At baseline, during the 1st trimester of pregnancy (gestational age (GA) up to 12 weeks +6 days)
  ICIQ-UI SF score between 0-21
Urinary incontinence at the 2nd trimester of pregnancy | At the follow-up at Gestational age 26 weeks and 0 days
  ICIQ-UI SF score between 0-21
Urinary incontinence incidence at the 3rd trimester of pregnancy | At the follow-up at Gestational Age 36 weeks and 0 days
  ICIQ-UI SF score between 0-21
Urinary incontinence incidence at 6 weeks postpartum | At the follow-up at 6 weeks postpartum
  ICIQ-UI SF score between 0-21
Anal incontinence (AI) incidence at inclusion, during the 1st trimester of pregnancy | At baseline, during the 1st trimester of pregnancy (gestational age (GA) up to 12 weeks +6 days)
  Colorectal-anal distress inventory 8 (CRAD-8), a part of Pelvic Floor Disability Index (PFDI-20) questionnaire: score calculated by the mean value of all item scores (possible 0-4) multiplied by 25 to obtain the score (range 0 to 100). Answer yes to one of the three questions about anal incontinence will be considered as AI.
Anal incontinence (AI) in the 2nd trimester of pregnancy | At the follow-up at Gestational Age 26 weeks and 0 days
  Colorectal-anal distress inventory 8 (CRAD-8), score 0-100. Answer yes to one of the three questions about anal incontinence will be considered as AI.
Anal incontinence (AI) incidence in the 3rd trimester of pregnancy | At the follow-up at Gestational Age 36 weeks and 0 days
  Colorectal-anal distress inventory 8 (CRAD-8), score 0-100. Answer yes to one of the three questions about anal incontinence will be considered as AI.
Anal incontinence (AI) incidence at 6 weeks postpartum | At the follow-up at 6 weeks postpartum
  Colorectal-anal distress inventory 8 (CRAD-8), score 0-100. Answer yes to one of the three questions about anal incontinence will be considered as AI.
Anal incontinence (AI) incidence at 3 months postpartum | At the follow-up at 3 months postpartum
  Colorectal-anal distress inventory 8 (CRAD-8), score 0-100. Answer yes to one of the three questions about anal incontinence will be considered as AI.
Anal incontinence (AI) incidence at 6 months postpartum | At the follow-up at 6 months postpartum
  Colorectal-anal distress inventory 8 (CRAD-8), score 0-100. Answer yes to one of the three questions about anal incontinence will be considered as AI.
Sexual dysfunction incidence at inclusion, during the 1st trimester of pregnancy | At baseline, during the 1st trimester of pregnancy (gestational age (GA) up to 12 weeks +6 days)
  Female Sexual Function Index-6 (FSFI-6) score between 2 to 30
Sexual dysfunction incidence at inclusion, during the 2nd trimester of pregnancy | At the follow-up at Gestational Age 26weeks and 0 days
  Female Sexual Function Index-6 (FSFI-6) score between 2 to 30
Sexual dysfunction incidence at inclusion, during the 3rd trimester of pregnancy | At the follow-up at Gestational Age 36 weeks and 0 days
  Female Sexual Function Index-6 (FSFI-6) score between 2 to 30
Sexual dysfunction incidence at 6 weeks postpartum | At the follow-up at 6 weeks postpartum
  Female Sexual Function Index-6 (FSFI-6) score between 2 to 30
Sexual dysfunction incidence at 3 month postpartum | At the follow-up at 3 month postpartum
  Female Sexual Function Index-6 (FSFI-6) score between 2 to 30
Sexual dysfunction incidence at 6month postpartum | At the follow-up at 6 month postpartum
  Female Sexual Function Index-6 (FSFI-6) score between 2 to 30
Pelvic organ prolapse (POP) incidence at inclusion, during the 1st trimester of pregnancy | At baseline, during the 1st trimester of pregnancy (gestational age (GA) up to 12 weeks and 6 days)
  Pelvic Organ Prolapse Distress Inventory 6 (POPDI-6), a part of Pelvic Floor Disability Index (PFDI-20) questionnaire: score calculated by the mean value of all item scores (possible 0-4) multiplied by 25 to obtain the score (range 0 to 100).
Pelvic organ prolapse (POP) incidence, in the 2nd trimester of pregnancy | At the follow-up at gestational age 26 weeks and 0 days
  Pelvic Organ Prolapse Distress Inventory 6 (POPDI-6), a part of Pelvic Floor Disability Index (PFDI-20) questionnaire: score calculated by the mean value of all item scores (possible 0-4) multiplied by 25 to obtain the score (range 0 to 100).
Pelvic organ prolapse (POP) incidence, in the 3rd trimester of pregnancy | At the follow-up at gestational age 36 weeks and 0 days
  Pelvic Organ Prolapse Distress Inventory 6 (POPDI-6), a part of Pelvic Floor Disability Index (PFDI-20) questionnaire: score calculated by the mean value of all item scores (possible 0-4) multiplied by 25 to obtain the score (range 0 to 100).
Pelvic organ prolapse (POP) incidence at 6 weeks postpartum | At the follow-up at 6 weeks postpartum
  Pelvic Organ Prolapse Distress Inventory 6 (POPDI-6), a part of Pelvic Floor Disability Index (PFDI-20) questionnaire: score calculated by the mean value of all item scores (possible 0-4) multiplied by 25 to obtain the score (range 0 to 100).
Pelvic organ prolapse (POP) incidence at 3 months postpartum | At the follow-up at 3 months postpartum
  Pelvic Organ Prolapse Distress Inventory 6 (POPDI-6), a part of Pelvic Floor Disability Index (PFDI-20) questionnaire: score calculated by the mean value of all item scores (possible 0-4) multiplied by 25 to obtain the score (range 0 to 100).
Pelvic organ prolapse (POP) incidence at 6 months postpartum | At the follow-up at 6 months postpartum
  Pelvic Organ Prolapse Distress Inventory 6 (POPDI-6), a part of Pelvic Floor Disability Index (PFDI-20) questionnaire: score calculated by the mean value of all item scores (possible 0-4) multiplied by 25 to obtain the score (range 0 to 100).
Length of the second stage of delivery | The outcome is registered in electronic patient journal during delivery, but the outcome will be collected during the first 3 months postpartum.
  Length in minutes (minimum 0 - maximum 300 minutes).
Delivery mode | The outcome is registered in electronic patient journal during delivery, but the outcome will be collected during the first 3 months postpartum.
  Vaginal, planned or unplanned Caesarean.
Foetal position | The outcome is registered in electronic patient journal during delivery, but the outcome will be collected during the first 3 months postpartum.
  Cephalic regular (occiput anterior), cephalic occiput posterior or breech
Episiotomy | The outcome is registered in electronic patient journal during delivery, but the outcome will be collected during the first 3 months postpartum
  Yes or no
Perineal tear | The outcome is registered in electronic patient journal during delivery, but the outcome will be collected during the first 3 months postpartum.
  Yes or no; if yes - tear degree (1st, 2nd, 3rd (3a, 3b, 3c), 4th)
Instrumental delivery | The outcome is registered in electronic patient journal during delivery, but the outcome will be collected during the first 3 months postpartum.
  Yes or no; if yes - type (vacuum assisted or forceps)
Length of the first stage of delivery | The outcome is registered in electronic patient journal during delivery, but the outcome will be collected during the first 3 months postpartum.
  Length in minutes (minimum 0 - no maximum)
Fidelity of PFMT | The questionnaire is filled every week from baseline to 6 months postpartum
  Self-reported training frequency (from 0 to 4 times a week)
Other implementation outcomes: acceptability, feasibility, appropriateness | At study completion
  Will be collected through short interviews

CONTACTS AND LOCATIONS:
Overall Officials: Jan Stener Jørgensen, Study Chair — University Hospital of Southern Denmark
Locations (1):
- Sygehus Sønderjylland, Aabenraa, Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No